CLINICAL TRIAL: NCT03898440
Title: Using Anogenital Distance to Determinate Fetal Gender Beetween 18 et 41 Weeks of Gestation.
Brief Title: Fetal Ano-genital Distance in 2D Ultrasound.
Acronym: DAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DAG (29BRC18.0067)
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-01

CONDITIONS: Urogenital Abnormalities; Prenatal Disorder; Sex Development Disorder
Keywords: anogenital distance; prenatal; sex determination; androgen
MeSH Terms: conditions — Urogenital Abnormalities; Disorders of Sex Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine a threshold value of fetal anogenital distance in 2D ultrasound to differentiate male fetuses from female fetuses, starting 18 weeks of gestation and until the due date.

The study also evaluates the feasibility of the measure and its interobserver variability.

DETAILED DESCRIPTION:
The anogenital distance of female newborns is shorter than that of male newborns.

Urogenital disorders, such as hypospadias and micro-penis, are associated with a shorter anogenital distance.

Anogenital distance is a good marker of fetal exposure to androgenic substances.

Prenatal anogenital distance ultrasound measure can help the diagnosis in case of doubt about fetal sexual phenotype or in case of urogenital disorder suspicion (hypospadias or micropenis).

Is the anogenital distance easy to make measure? Can this procedure be reproduced? What are the threshold values to determine fetal sex at each term of pregnancy?

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman
* sonographic fetal follow up in Brest Hospital
* term>18 weeks of gestation

Exclusion Criteria:

* No datation between 11 weeks of gestation and 13 weeks of gestation and 6 days by crown-rump length measurement
* Minor
* no consent
* ultrasound performed by an operator without ultrasonography graduation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All pregnant women follow up at Brest Hospital to 18 weeks of gestation until term, except suspicion of fetal pelvic malformations and patients without an exact echographic datation of pregnancy between 11 and 13+6 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
fetal anogenital distance | During fetal ultrasound exam
  The distance will be measured from the center of the anus to the posterior convergence of the fourchette in female fetuses and to the posterior base of the scrotum in male fetuses

SECONDARY OUTCOMES:
Interobserver variability | During fetal ultrasound exam
  reproducibility of the anogenital measure: the measure will be taken by two sonographers during the same exam
Ano-genital distance in mm | During fetal ultrasound exam
  the measure is correctly performed and validated by an expert
Estimated fetal weight | During fetal ultrasound exam
  Impact of estimated fetal weight and anogenital distance
neonatal sex determination | During fetal ultrasound exam
  concordance of anogenital distance and neonatal sex determination

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Hélène SALIOU, Principal Investigator — CHRU Brest - Morvan hospital
Locations (1):
- CHRU de Brest (Morvan), Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement